CLINICAL TRIAL: NCT02449057
Title: An Evaluation of JUST (Juveniles Under Supervision and Treatment) Court in Yuma County, AZ
Brief Title: An Evaluation of JUST Court in Yuma County, AZ
Acronym: JUST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pepperdine University (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SPP1014F01
Record Dates: First submitted 2015-02-10; First posted 2015-05-20 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Substance Abuse; Adolescent Behavior; Juvenile Delinquency Unspecified
MeSH Terms: conditions — Substance-Related Disorders; Adolescent Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- JUST (Experimental): Juveniles Under Supervision and Treatment. This entails swift, certain, and modest sanctions for violations of terms of community supervision.
  Interventions: Other: JUST
- Probation-as-Usual (No Intervention): Juvenile probation-as-usual.

INTERVENTIONS:
Other: JUST — Swift, certain, and proportionate sanctions for violations of terms of community supervision.
  Arms: JUST

SUMMARY:
Arizona has created a pilot program for juvenile probationers called Juveniles under Supervision and Treatment (JUST), which includes swift and certain, but modest responses, to technical violations of the terms of juvenile probation. JUST targets high- and medium-risk juvenile probationers and its stated objective is to reduce violations and overall incarceration of youth in the program. The JUST pilot is being implemented under the authority of the Arizona Governor's Office for Children, Youth and Families (GOCYF) and the Administrative Office of the Courts (AOC).

DETAILED DESCRIPTION:
Arizona's Juveniles Under Supervision and Treatment (JUST) Court is a pilot project initiated by the Arizona Governor's office. It is designed to test whether the principles of Swift, Certain, and Fair (SCF) Supervision-clear rules, close monitoring, and swift and certain, but modest, penalties for each violation can succeed when applied to juveniles under community supervision. The Arizona Administrative Office of the Courts piloted JUST in two counties: Yavapai and Yuma. The Yuma program was launched in March 2011. The goal of JUST is to (a) reduce the violation rate so as to reduce the number of petitions filed to revoke probation (the purpose is to reduce the use of juvenile detention), and (b) reduce recidivism overall. All juveniles in Yavapai are supervised under JUST (evaluation using an RCT is therefore unfeasible). JUST in Yuma is now being scaled up, which affords the opportunity for an RCT. The goal of the RCT is to compare the performance of youth supervised under JUST with those supervised under probation-as-usual.

ELIGIBILITY:
Inclusion Criteria:

* Newly probated
* At least 13 years old
* No older than 17 years and 3 months
* At least nine months remaining on supervision
* Must be on standard probation with a supervision level of moderate to maximum
* Must be able to participate in the program for at least nine months

Exclusion Criteria:

* Not meeting all inclusion criteria
* Sex offender
* Dangerous offenses

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Number of days served in detention | followup at 6 months
  Number of days served in detention
Recidivism | followup at 6 months
  Number of new arrests (overall, and by type)

SECONDARY OUTCOMES:
Truancy | followup at 6 months
  Number of days truant
Failure to appear | followup at 6 months
  Number of no-shows for probation appointments
Other technical violations | followup at 6 months
  Number of other technical violations
Substance use | followup at 6 months
  Results of urinalysis screens from routine testing and research-based testing
New dispositions | followup at 6 months
  Number of new dispositions, by (type)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Hawken, PhD, Principal Investigator — Pepperdine University
Locations (1):
- Yuma County Juvenile Justice Center, Yuma, Arizona, United States